CLINICAL TRIAL: NCT02753426
Title: A Trial of Doxycycline in Renal Disease (ADORE)
Brief Title: A Trial of Doxycycline in Renal Disease
Acronym: ADORE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 15-17569
Record Dates: First submitted 2016-04-24; First posted 2016-04-27 (Estimated); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: Chronic Kidney Disease; Cardiorenal Syndrome
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardio-Renal Syndrome | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Doxycycline-Placebo (Other): Doxycycline 20mg capsule for 30 days, 30-day washout, and then placebo capsule for 30 days.
  Interventions: Drug: Doxycycline; Drug: Placebo (for Doxycycline)
- Placebo-Doxycycline (Other): Placebo capsule for 30 days, 30-day washout, and then Doxycycline 20mg capsule for 30 days.
  Interventions: Drug: Doxycycline; Drug: Placebo (for Doxycycline)

INTERVENTIONS:
Drug: Doxycycline — Doxycycline 20mg capsule by mouth, twice a day for 30 days.
Drug: Placebo (for Doxycycline) — Inactive pill manufactured to mimic Doxycycline 20mg. Capsule by mouth, twice a for 30 days.

SUMMARY:
The goal of this trial is to evaluate whether subantimicrobial-dose of doxycycline (20mgBID) will affect serum and urine biomarkers of fibrosis in patients with pre-dialysis chronic kidney disease.

DETAILED DESCRIPTION:
This is a Phase I, placebo-controlled, randomized crossover trial to determine the effects of 4-week treatment with subantimicrobial-dose doxycycline on serum and urine biomarkers of fibrosis in patients with pre-dialysis chronic kidney disease (eGFR<30ml/min/1.73m2). Doxycycline is a matrix metalloproteinase inhibitor and is approved for use as an anti-fibrotic in the setting of gum and skin disease at low doses (20mgBID). At such a dose, serum levels are too low for antimicrobial effect and chronic usage is not thought to lead to tetracycline resistance. Investigators hypothesize that doxycycline will ameliorate cardiac and renal fibrosis and thus investigators will detect a decrease in fibrotic markers during treatment with doxycycline.

ELIGIBILITY:
Inclusion Criteria:

* CKD pre-dialysis (eGFR< 30 ml/min/1.73m2 not on dialysis);
* local 415/650/510 area codes;
* primary language English or Spanish

Exclusion Criteria:

* eGFR worsening by greater than 5ml/min/1.73 m2 during the last 6 months;
* Systolic blood pressure less than 100mmHg or greater than 170 mmHg;
* pregnancy;
* ejection fraction less than 45%;
* NYHA class III or IV HF;
* myocardial infarction or hospitalization for HF within 4 months;
* liver disease;
* moderate or severe chronic obstructive pulmonary disease or pulmonary fibrosis;
* current infection;
* chemotherapy;
* major surgery within last month;
* bilateral dialysis access precluding lab draw;
* self-reported use of IV drugs or cocaine within the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-04; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Serum markers of fibrosis | 3 months
  Serum collagen type III amino-terminal propeptide (PIIINP), soluble suppression of tumorigenicity 2 (ST2)
Urinary markers of fibrosis | 3 months
  Urinary PIIINP, Urinary alpha-1 macroglobulin (A1M)

SECONDARY OUTCOMES:
Adverse effects | 3 months
  Nausea, rash

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Dubin, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No